CLINICAL TRIAL: NCT05622253
Title: Combined Low-Dose Isotretenion and Long-Pulsed 1064 ND-YAG Laser in the Treatment of Acne Erythema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Essam, Lecturer of Dermatology, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5566-RE
Record Dates: First submitted 2022-11-12; First posted 2022-11-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Low-Dose Isotretenion and Long-Pulsed 1064 ND-YAG Laser in the Treatment of Acne Erythema (Experimental): Selected patients will be treated with low-dose oral isotretinoin (10mg/day) over a period of sessions and six sessions of 1064 ND- YAG laser (Deka motous AY) using 150 J/cm2, 20-25 milliseconds pulse duration, and 5 mm spot size, at 2 weeks' interval.
  Interventions: Combination Product: Combined Low-Dose Isotretenion and Long-Pulsed 1064 ND-YAG Laser

INTERVENTIONS:
Combination Product: Combined Low-Dose Isotretenion and Long-Pulsed 1064 ND-YAG Laser — Selected patients will be treated with low-dose oral isotretinoin (10mg/day) over a period of sessions and six sessions of 1064 ND- YAG laser (Deka motous AY) using 150 J/cm2, 20-25 milliseconds pulse duration, and 5 mm spot size, at 2 weeks' interval.

SUMMARY:
Acne erythema consists of telangiectasia and erythematous papules, without a comedo, which occurs as a result of inflammatory acne. Moreover, although acne erythema is common in acne patients, no satisfactory medical or surgical treatment is available for this condition. Some acne erythema lesions may improve with time, but the persistent acne erythema, which is experienced by most patients, is cosmetically unacceptable and leads to frustration and psychological distress.

DETAILED DESCRIPTION:
Up to the present time, there have been several studies on the clinical efficacy of different laser modalities for acne treatment. Pulsed dye laser (PDL), 585 or 595 nm, has been demonstrated as one of the effective treatment options Another laser long-pulsed neodymium: yttrium-aluminum-garnet (Nd:YAG) laser with 1064 nm has been commonly used for skin rejuvenation. Nevertheless, the efficacy of this laser for acne treatment has been shown in some studies and case reports. The therapeutic effect on acne lesions is believed to be mediated by the selective photothermolysis of vessels, the upregulation of TGF-β, the reduction of interleukin-8 (IL-8) and Toll-like receptors-2 (TLR-2), and the thermal destruction of sebaceous glands.

Isotretinoin remains the mainstay of acne treatment. No doubt, the side effects of this effective drug holds physicians back from jumping to prescribe it. Recent data suggested that lower doses (0.25 mg/kg/day) may lead to fewer side effects. and fewer flares. Clearing the use of oral isotretinoin in combination with other procedures has expanded our therapeutic options to obtain better control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult Patients with acne 2. Patients of both sexes. 3. Willing to sign an informed consent

Exclusion Criteria:

- 1. Patients who were taking concomitant acne medication 2. Patients had a history of topical or systemic therapy use for acne for the past 6 months, 3. Patients with a history of photosensitivity reactions 4. Patients with any renal or hepatic compromise or any preexisting hyperlipidemia.

5. Pregnant females as well as females who intend to become pregnant during treatment 6. Hypertrophic scar or keloid. 7. Active or recurrent herpes simplex.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The degree of acne erythema was determined on the 4-point grading of acne erythema | 4 months
  0 None Clear
  1. Mild Faintly detectable erythema, light pink
  2. Moderate Dull red, clearly distinguishable
  3. severe Deep/dark red

CONTACTS AND LOCATIONS:
Overall Officials: Reham Essam, MD, Principal Investigator — Zagazig University
Locations (1):
- Reham Essam, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: No